CLINICAL TRIAL: NCT01342809
Title: Follow up After Self-poisoning by General Practitioner- a Randomised Clinical Trial
Brief Title: Follow up by General Practitioner After Self-poisoning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Lovisenberg Diakonale Hospital (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Tine K. Grimholt, Phd candidate, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-08708b
Record Dates: First submitted 2011-04-18; First posted 2011-04-27 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Suicidal and Self-injurious Behaviour
Keywords: Depression; Hopelessness; Suicidal ideation
MeSH Terms: conditions — Self-Injurious Behavior; Depression; Suicidal Ideation | interventions — General Practitioners

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow up (Experimental): Close follow up from written guidelines, supervision provided.
  Interventions: Behavioral: Follow up
- Usual Treatment (No Intervention)

INTERVENTIONS:
Behavioral: Follow up — Follow up, consultations with general practitioner, written guidelines, supervision.
  Other Names: General Practitioner
  Arms: Follow up

SUMMARY:
The study hypothesis is that follow up from general practitioner after hospitalization for self poisoning will decrease suicidal behaviour.

DETAILED DESCRIPTION:
Patients hospitalized after an episode of self poisoning will be randomly assigned into intervention an control groups. The intervention is close follow up by general practitioner six months. Both groups will receive treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Self Poisoning (according to the WHO definition)
* Ability to fill out questionnaire

Exclusion Criteria:

* Hospitalization into psychiatric ward
* Unknown address or ID
* Not registered with General Practitioner
* If institutionalized or in jail.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-11; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Suicidal behaviour | 3 and 6 months
  Beck Cepression Inventory, Beck Hopelessness scale, Beck Suicide Ideation Scale
Suicidal behaviour | 3 and 6 months
  Beck Depression Inventory, Beck Hopelessness scale, Beck Suicide Ideation Scale

SECONDARY OUTCOMES:
Treatment | 3 and 6 months
  Contacts with GP, and health care services, satisfaction with treatment GP (EUROPEP)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Grimholt TK, Jacobsen D, Haavet OR, Sandvik L, Jorgensen T, Norheim AB, Ekeberg O. Effect of Systematic Follow-Up by General Practitioners after Deliberate Self-Poisoning: A Randomised Controlled Trial. PLoS One. 2015 Dec 2;10(12):e0143934. doi: 10.1371/journal.pone.0143934. eCollection 2015. PMID 26629812
- [Derived] Grimholt TK, Jacobsen D, Haavet OR, Sandvik L, Jorgensen T, Norheim AB, Ekeberg O. Structured follow-up by general practitioners after deliberate self-poisoning: a randomised controlled trial. BMC Psychiatry. 2015 Oct 14;15:245. doi: 10.1186/s12888-015-0635-2. PMID 26467530